CLINICAL TRIAL: NCT06425354
Title: Use of 'Mechanical Power' as a Predictor of Increased Serum and Pulmonary Proinflammatory Cytokine Concentrations in Patients With Acute Hypoxemic Respiratory Failure: A Prospective Observational Study
Status: Recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Alessandri, Prof, University of Roma La Sapienza
Other Study IDs: RIA24.1
Record Dates: First submitted 2024-05-17; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Mechanical Power
MeSH Terms: interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma serum and BAL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mechanical ventilation — Mechanical ventilatiom

SUMMARY:
The aim of this study is to report the proportion of patients with acute hypoxemic respiratory failyre (AHRF) undergoing mechanical ventilation who exceed 17 J/min of mechanical power (MP) and the difference in terms of proinflammatory cytokine concentration in blood samples and bronchoalveolar lavage.

The main questions it aims to answer are:

1. Which is the proportion of patients who exceed 17 J/min of mechanical power (MP) during the first 72 hours of mechanical ventilation?
2. Is there a difference in terms of cytokine concentration in patients undergoing mechanical power >17 J/min compared to <17 J/min?

Patients will be divided into two groups based on respiratory mechanics measurements: low MP group (average MP <17 J/min) and high MP group (average MP ≥17 J/min). The researchers will collect blood and BAL samples and perform cytokine assays.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AHRF (P/F <300 mmHg) undergoing invasive mechanical ventilation within 7 days from the onset of symptoms
* Invasive mechanical ventilation for less than 6 hours
* Evidence of newly developed lung consolidation on chest imaging (X-ray, CT)
* Age ≥18 years

Exclusion Criteria:

* Prior invasive mechanical ventilation during the same hospitalization
* Tracheostomy
* Severe anemia (Hb<7g/dL)
* Severe neutropenia
* Renal insufficiency or RRT (Renal Replacement Therapy)
* Noradrenaline >0.5 mcg/kg/min
* Pregnancy
* Extracorporeal circulation (ECCO2R, ECMO)
* Life expectancy <24 hours as clinically judged
* Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AHRF undergoing mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Patients who exceed 17 J/min of MP | 4 years
  Proportion of patients with AHRF undergoing mechanical ventilation who exceed 17 J/min of MP

SECONDARY OUTCOMES:
Inflammatory cytokines | 4 years
  Difference in terms of proinflammatory cytokine concentration in blood samples and bronchoalveolar lavage.

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided